CLINICAL TRIAL: NCT06238024
Title: Effect of Interleukin-6 Receptor Inhibition in Patients With Ischemic Stroke Undergoing Endovascular Treatment: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Effect of Interleukin-6 Receptor Inhibition in Patients With Ischemic Stroke Undergoing Endovascular Treatment
Acronym: IRIS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Suzhou Municipal Hospital of Anhui Province (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZSLYY
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-07

CONDITIONS: Interleukin-6; Ischemic Stroke; Endovascular Treatment
Keywords: Acute ischemic stroke; Tocilizumab; Neuroprotection; Outcome
MeSH Terms: conditions — Ischemic Stroke | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab group (Experimental): Intravenously for more than 1 hour.
  Interventions: Drug: Tocilizumab
- Control group (Placebo Comparator): Intravenously for more than 1 hour.
  Interventions: Drug: NaCl 0.9% 100ml

INTERVENTIONS:
Drug: Tocilizumab — Single dose intravenous application
  Arms: Tocilizumab group
Drug: NaCl 0.9% 100ml — Single dose intravenous application
  Arms: Control group

SUMMARY:
Tocilizumab may exert neuroprotective effects in patients with ischemic stroke undergoing endovascular treatment

DETAILED DESCRIPTION:
Vascular recanalization techniques, including thrombolysis and thrombectomy, have become the mainstay of treatment for acute ischemic stroke. However, some patients still experience poor prognosis, with ineffective recanalization and reperfusion brain injury being the major contributors to unfavorable outcomes. Studies have indicated that tocilizumab, used in ST-segment elevation and non-ST-segment elevation myocardial infarction, exhibits anti-inflammatory and myocardial protective effects. Nevertheless, whether tocilizumab can provide neuroprotection in the early stages of acute large vessel recanalization remains uncertain. Given the above evidence, the aim of this study was to investigate whether combination therapy with tocilizumab in the early phase of recanalization of acute large vessel occlusion could further exert a beneficial effect and thus improve the poor prognosis of patients.

ELIGIBILITY:
* Inclusion criteria:

  1. Age 18-80 years.
  2. Acute ischemic stroke caused by occlusion of intracranial segment of the internal carotid artery, middle cerebral artery M1, or M2 segment.
  3. NIHSS ≥ 6.
  4. Meeting the criteria of endovascular treatment:

     ① ASPECTS score ≥ 6, possibile to start endovascular treatment within 6 hours from stroke onset.

     ② Stroke onset between 6-16 hours, meeting DEFUSE-3 criteria (infarct core volume < 70ml, mismatch ratio ≥ 1.8, and mismatch volume > 15ml), or DAWN criteria (NIHSS ≥ 10 and infarct core volume < 31ml; or NIHSS ≥ 20 and infarct volume 31-51ml).

     ③ Stroke onset between 16-24 hours, meeting DAWN criteria (NIHSS ≥ 10 and infarct core volume < 31ml; or NIHSS ≥ 20 and infarct volume 31-51ml).

     ④ When ASPECTS score is < 6, meeting RESCUE-Japan LIMIT criteria (ASPECTS score 3-5; stroke onset within 6 hours or between 6-24 hours but no acute stroke signs on FLAIR), or ANGEL-ASPECT criteria (stroke onset within 24 hours, ASPECTS 3-5; or onset within 24 hours, ASPECTS 0-2 and infarct core volume 70-100 mL; or onset between 6-24 hours, ASPECTS > 5 and infarct core volume 70-100 mL), or SELECT2 criteria (ASPECTS 3-5; or infarct core volume greater than 50ml).
  5. Experimental drug administration had to be possible within 24 hours after stroke onset.
  6. Obtained Informed consent from the patient or their legal representative.
* Exclusion Criteria:

  1. Hemorrhagic diseases visible on head CT: hemorrhagic stroke, epidural hematoma, subdural hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc.
  2. Pre-stroke mRS score > 1.
  3. Known allergy to tocilizumab or excipients.
  4. Known allergy to iodinated contrast agents.
  5. Anticipated difficulty in completing endovascular treatment due to vascular tortuosity.
  6. History of congenital or acquired bleeding disorders, coagulation factor deficiency diseases, thrombocytopenic diseases, etc.
  7. Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg despite blood pressure control.
  8. Neutrophil < 2×10 9/L.
  9. Platelet < 100×10 9/L.
  10. Blood glucose < 2.8 mmol/L (50 mg/dl) or > 22.2 mmol/L (400 mg/dl).
  11. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 1.5 times the upper limit of normal.
  12. Known recent or current serum creatinine exceeding 1.5 times the upper limit of normal or estimated glomerular filtration rate (eGFR) < 60 mL/min.
  13. Pregnant, lactating, or planning pregnancy within 90 days.
  14. Severe mental disorders or inability to comply with informed consent and follow-up requirements due to dementia.
  15. Concurrent malignant tumors or severe systemic diseases with an expected survival of less than 90 days.
  16. Presence of autoimmune diseases or use of immunosuppressive drugs.
  17. Systemic infectious diseases
  18. Participation in another interventional clinical study within 30 days before randomization or currently participating in another interventional clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-09-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in infarct-core volume | 72 hours
  The infarct-core volume is determined by diffusion-weighted MRI, CT, or CTP images.

SECONDARY OUTCOMES:
Early neurological improvement | within 24 hours
  Decrease in National Institute of Health stroke scale (NIHSS) score of ≥8 or NIHSS score of 0-2 within 24 hours. NIHSS scores range from 0 to 42, with higher scores indicating greater neurologic deficit
NIHSS score | 24 hours
  National Institutes of Health Stroke Scale (NIHSS) scores range from 0 to 42, with higher scores indicating greater neurologic deficit
Proportion of successful reperfusion (mTICI 2b/3) | immediate postoperative
  mTICI denotes modified Treatment in Cerebral Ischemia classification, with scores ranging from 0 (no flow) to 3 (normal flow)
Proportion of recanalization on follow-up CTA or MRA | 72 hours
Incidence of cerebral hemorrhage | 72 hours
Incidence of symptomatic cerebral hemorrhage | 72 hours
NIHSS score | 7 days
  National Institutes of Health Stroke Scale (NIHSS) scores range from 0 to 42, with higher scores indicating greater neurologic deficit
Incidence of stroke-associated pneumonia | 7 days
Incidence of decompressive craniectomy | 7 days
Proportion of patients with functional independence (mRS 0-2) | 90 days
  Scores on the modified Rankin scale range from 0 to 6, with higher scores indicating greater disability
Shift analysis of mRS score | 90 days
  Scores on the modified Rankin scale range from 0 to 6, with higher scores indicating greater disability
Barthel Index | 90 days
  The Barthel index is an ordinal scale for measuring performance of activities of daily living. Scores ranges from 0 to 20, with 0 indicating severe disability and 19 or 20 indicating no disability that interferes with daily activities.
EuroQoL Group 5-Dimension Self-Report Questionnaire (EQ-5D) | 90 days
  EQ-5D is a standardized instrument for the measurement of health status. Scores range from -0.33 to 1.00, with higher scores indicating a better quality of life
Death | 90 days
Adverse events and serious adverse events | 90 days

OTHER OUTCOMES:
Change of hsCRP levels from admission to 72 hours | 72 hours
Change of inflammatory blood biomarkers | baseline, 24 hours, 48 hours, and 72 hours
  Interleukin-6

CONTACTS AND LOCATIONS:
Overall Officials: Chuanjie Wu, M.D., Study Director — Xuanwu Hospital, Beijing; Zhengfei Ma, M.M., Study Director — Suzhou Municipal Hospital of Anhui Province; Xunming Ji, M.D., Study Chair — Xuanwu Hospital, Beijing; Xuehong Chu, M.D., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Suzhou Municipal Hospital of Anhui Province, Suzhou, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes